CLINICAL TRIAL: NCT06978699
Title: A Multicenter, Randomized, Single-blind Phase II Study Evaluating the Efficacy and Safety of XH-S003 Capsules in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Brief Title: A Phase II Study Evaluating the Efficacy and Safety of XH-S003 Capsules in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Acronym: XH-S003-II-101
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: S-INFINITY Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XH-S003-II-101
Record Dates: First submitted 2025-05-08; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: PNH - Paroxysmal Nocturnal Hemoglobinuria
Keywords: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose 1 (Experimental): Once daily
  Interventions: Drug: XH-S003 Capsule
- Dose 2 (Experimental): Once daily
  Interventions: Drug: XH-S003 Capsule
- Dose 3 (Experimental): Once daily
  Interventions: Drug: XH-S003 Capsule

INTERVENTIONS:
Drug: XH-S003 Capsule — 25mg & 100mg

SUMMARY:
This is a multicenter, randomized, single-blind Phase II trial to evaluate the efficacy and safety of XH-S003 capsules in PNH patients. About 24 PNH patients will be enrolled and randomized to three dose levels and take XH-S003 capsules orally

ELIGIBILITY:
Inclusion Criteria:

* Male or female with aged ≥18 years old;
* Weight ≥40 kg and BMI≥18 kg/m2 ;
* Diagnosed with PNH: with red blood cell or granulocyte clone levels >10% detected by flow cytopy within 6 months prior to screening or during screening;
* Patients who have not previously received any complement inhibitor therayp;
* LDH > 1.5×ULN detected two times during the screening period (interval of 2 to 8 weeks);
* Hb meets one of the following conditions: (1) Hb <100 g/L at the first screening visit, and subjects receive RBC transfusion because of PNH-related anemia during the screening period; (2) The average Hb of two tests during the screening period <100 g/L (interval of 2~8 weeks);
* Vaccination against Neisseria meningitidis and Streptococcus pneumoniae before the first administration. If the subject has not been vaccinated previously or requires booster vaccination (according to local vaccination policies), vaccination must be administered at least 2 weeks before the first administration. If the first administration must begin less than 2 weeks after vaccination, preventive antibiotic treatment must begin at least 2 weeks after vaccination;

Exclusion Criteria:

* Subjects with laboratory evidence of bone marrow failure during the screening period (reticulocyte count <100×109/L, platelet count <30×109/L, or neutrophil count <0.5×109/L);
* Subjects receiving other therapies prior to screening who have not achieved the following treatment durations:

  • Erythropoietin or immunosuppressants for at least 8 weeks; • Systemic corticosteroids for at least 4 weeks; • Iron supplements, vitamin B12, or folic acid for at least 4 weeks; • Anticoagulants: Vitamin K antagonists for at least 4 weeks with stable international normalized ratio (INR) (as determined by the investigator), low molecular weight heparin for at least 4 weeks; • Hypoxic-inducing factor prolyl hydroxylase inhibitors (HIF-PHI) for at least 8 weeks; • Androgens for at least 4 weeks;
* A history of bone marrow/hematopoietic stem cell or solid organ transplantation;
* Alanine aminotransferase (ALT), γ-glutamyl transpeptidase (GGT), or alkaline phosphatase (ALP) >3×ULN at screening; - Positive HIV antibody, active syphilis infection, positive HBsAg, active HCV infection, or active tuberculosis infection at screening;
* Known or suspected immunodeficiency diseases or hereditary complement deficiency at screening;
* A history of Neisseria meningitidis infection;
* Subjects with chronic active or recurrent infections within 1 year prior to screening;
* Subjects with systemic active bacterial, viral (including COVID-19), or fungal infections within 2 weeks prior to the first administration; subjects with body temperature >38°C within 7 days prior to the first administration;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological sex of eligible participants.
Enrollment: 24 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Changes of hemoglobin compared with baseline | 8 weeks
  Changes of hemoglobin compared with baseline

SECONDARY OUTCOMES:
Proportion of subjects with an increase in Hb ≥20g/L compared with baseline (without RBC transfusion); | 8 weeks
  Proportion of subjects with an increase in Hb ≥20g/L compared with baseline (without RBC transfusion);
Changes in Indirect Bilirubin compared to baseline; | 8 weeks
  Changes in Indirect Bilirubin compared to baseline;
Changes in reticulocyte counts compared to baseline; | 8 weeks
  Changes in reticulocyte counts compared to baseline;
Proportion of subjects without RBC transfusion | 8 weeks
  Proportion of subjects without RBC transfusion
Changes in LDH compared with baseline | 8 weeks
  Changes in LDH compared with baseline

CONTACTS AND LOCATIONS:
Locations (1):
- TianJin Medical University General Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No